CLINICAL TRIAL: NCT00241098
Title: A Randomized, Double Blind, Parallel Group Study to Evaluate the Effects of Valsartan Versus Placebo in Patients With Early Stage Heart Failure Due to Diastolic Dysfunction Already Evidenced by an Elevated B-type Natriuretic Peptide Level: the VALIDATE Study
Brief Title: The VALIDATE Study of Valsartan for Patients With Early Stage Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489B2402
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Hypertension; Congestive Heart Failure
Keywords: HYPERTENSION; HEART FAILURE; PEPTIDE; valsartan
MeSH Terms: conditions — Hypertension; Heart Failure | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
This is a study to evaluate the response of patients with hypertension and early stage heart failure to valsartan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 25-85 years of age, inclusive
* Past diagnosis of hypertension for a min 1 year
* Patients with an established treatment regimen for hypertension with one or more agents for a minimum period of 2 months
* BP is considered adequately controlled with DBP < 90mmHg
* Elevated BNP levels both in bedside test (62pg/ml) and after validation of a separate blood sample (40pg/ml) in the central laboratory
* LV ejection fraction ³ 45%
* LVH defined as myocardial mass ³ 116 g /m2 in males and 104 g/m2 in females
* At least one of the following parameters of diastolic dysfunction

  * E/A < 1 for the patients who are younger than 55 years or < 0.8 for the patients whose age is ³ 55 years (full year), or
  * DT > 220 ms, or
  * IVRT > 90 ms

Exclusion Criteria:

• Present use of ACE inhibitor

Other protocol-defined exclusion criteria may apply.

-

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2003-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in a blood measurement for heart failure after 26 weeks

SECONDARY OUTCOMES:
Change from baseline in a blood measurement for heart failure after 12 weeks
Change in baseline heart size after 26 weeks
Change in baseline heart size, heart function, and other parameters of diastolic heart dysfunction after 26 weeks
Change from baseline in markers of heart fibrosis after 26 weeks
Change from baseline quality of life questionnaire after 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical, Study Director — Novartis Pharmaceuticals